CLINICAL TRIAL: NCT05151003
Title: Analysis of In-hospital Acute Kidney Injury Epidemiology, Treatment and Outcomes
Brief Title: Epidemiology of In-hospital Acute Kidney Injury
Acronym: GENAKI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universita degli Studi di Genova (Other)
Collaborators: Ospedale Policlinico San Martino (Other)
Responsible Party: Principal Investigator, Pasquale Esposito, Professor of Nephrology, Universita degli Studi di Genova
Other Study IDs: CER Liguria: 515/2020
Record Dates: First submitted 2021-11-15; First posted 2021-12-09 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Acute Kidney Injury; Dialysis; Complications; Chronic Kidney Diseases
MeSH Terms: conditions — Acute Kidney Injury; Renal Insufficiency, Chronic | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients admitted to University Hospital San Martino, Genova, Italy: Adult patients admitted to University Hospital San Martino, Genova, Italy
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Collection and analysis of data related to AKI epidemiology, treatment and outcomes

SUMMARY:
Retrospective observational study to investigate acute kidney injury (AKI) epidemiology and outcomes in patients hospitalized in University Hospital San Martino, Genova, Italy.

DETAILED DESCRIPTION:
A retrospective observational study was designed to investigate acute kidney injury (AKI) epidemiology and outcome in patients hospitalized in University Hospital San Martino, Genova, Italy.

All data will be extracted from the hospital electronic database. The investigators will evaluate demographic, clinical and laboratory data, including age, sex, serum creatinine (sCr), sodium and electrolytes, intensive care unit (ICU) admission, length of hospital stay, death, comorbidities and primary diagnosis codes at the hospital discharge (using International Classification of Diseases-ICD-9- codes).

The investigators will include also patients affected by Coronavirus disease 19 (COVID-19).

The primary endpoint will be to describe AKI epidemiology, secondary endpoints will be to evaluate AKI-related risk factors and clinical outcomes, such as length of stay and mortality.

Moreover, the investigators will describe the differences in the outcome and treatments of AKI patients in the medical wards and ICU.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to University Hospital San Martino, Italy
* We'll include also patients affected by Coronavirus disease 19 (COVID-19).

Exclusion Criteria:

* Hemodialysis patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to Policlinico Universitario San Martino, Genova, Italy (including those with COVID-19).
Sampling Method: Non-Probability Sample
Enrollment: 60000 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Acute Kidney Injury incidence | Collection of retrospective data from 2016
  Rate of in-hospital Acute Kidney Injury incidence
Acute Kidney Injury severity | Collection of retrospective data from 2016
  Staging of in-hospital Acute Kidney Injury according to the KDIGO guidelines

SECONDARY OUTCOMES:
Mortality in Acute Kidney Injury patients | Collection of retrospective data from 2016
  Rate of in-hospital mortality among patients with Acute Kidney Injury
Creatinine clearance after discharge | Collection of retrospective data from 2016
  Data on kidney function after the discharge in Acute Kidney Injury patients

CONTACTS AND LOCATIONS:
Overall Officials: Pasquale Esposito, Prof, Principal Investigator — University of Genova, Italy
Locations (1):
- IRCCS Policlinico San Martino, Genova, Italy

IPD SHARING:
Plan to Share IPD: No
Patient data will be anonymized.